CLINICAL TRIAL: NCT07271303
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Efficacy and Safety of Hyoscine Butylbromide Capsules for Preoperative Preparation in Painless Gastrointestinal Endoscopy Procedures
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of Hyoscine Butylbromide Capsules for Preoperative Preparation in Painless Gastrointestinal Endoscopy Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaobo Li, Chief physician, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: LY2025-335-A
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Painless Gastrointestinal Endoscopy
Keywords: Painless gastrointestinal endoscopy; Hyoscine Butylbromide; Preoperative Preparation
MeSH Terms: interventions — Butylscopolammonium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyoscine Butylbromide Group (Experimental): Participants receive hyoscine butylbromide capsules orally before painless gastrointestinal endoscopy
  Interventions: Drug: Hyoscine Butylbromide
- Placebo group (No Intervention): Participants receive matching placebo capsules orally before painless gastrointestinal endoscopy

INTERVENTIONS:
Drug: Hyoscine Butylbromide — Participants receive hyoscine butylbromide capsules orally before painless gastrointestinal endoscopy
  Arms: Hyoscine Butylbromide Group

SUMMARY:
Gastrointestinal endoscopy procedures, including upper gastrointestinal endoscopy and colorectal endoscopy, represent a fundamental and important method for examining and managing digestive tract diseases, with both diagnostic and therapeutic applications. They are also utilized as effective tools for surveillance of gastrointestinal tumors. During upper gastrointestinal endoscopy procedures, gastric peristalsis may restrict the operative field of view and access, significantly affecting procedural precision. Excessive peristalsis not only affects the observation of simple lesions but also impacts other procedural maneuvers Therefore, during upper gastrointestinal endoscopy procedures, antispasmodic agents are commonly used to suppress gastrointestinal motility, ultimately facilitating endoscopic visualization. However, most antispasmodic agents, such as hyoscine butylbromide (Buscopan), cimetropium bromide (Algiron), and atropine, must be administered by injection. Intravenous or intramuscular administration causes patient pain and anxiety, and increases medical costs. Some researchers have taken an alternative approach by spraying L-menthol onto the gastric mucosa during gastroscopy to reduce gastric peristalsis. Although study results and adverse reaction profiles have demonstrated its superiority, the application process still presents operational inconveniences. Furthermore, these drugs should be used with caution as they may cause potential adverse reactions, including dry mouth, urinary retention, temporary impairment of visual accommodation, palpitations, anaphylactic shock, and hyperglycemia.

DETAILED DESCRIPTION:
Here is the English translation for your study procedures:

1. Screening Period (Day -7 to Day -1) The following procedures or assessments are required during the screening period. Electrocardiogram results obtained within 7 days prior to randomization are acceptable. Blood biochemistry, complete blood count, and blood (urine) pregnancy test results obtained within 7 days prior to randomization are acceptable, including results completed before signing informed consent.

   Signing of informed consent form; Demographics and medical history collection; medical history is limited to current comorbidities and does not include conditions that have been cured; Vital signs: temperature, pulse, blood pressure; Physical examination: general condition, skin and mucosa, head and neck, chest, abdomen; 12-lead electrocardiogram; Complete blood count including at least: red blood cell count, white blood cell count, hemoglobin, platelet count; Blood biochemistry including at least: total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), creatinine, urea/blood urea nitrogen (BUN); Blood (urine) pregnancy test; Verification of inclusion/exclusion criteria.
2. Randomization and Blinding This study employs a random number table method, using SAS version 9.4 or above or other software for randomization. A randomization code table for no fewer than 74 subjects will be generated with a 1:1 ratio between the treatment group and control group. The study is double-blind; hyoscine butylbromide capsules and placebo are identical in appearance, packaging, and administration method, so that neither investigators nor subjects can determine group assignment based on the medication itself. Medications will be dispensed by an independent third party (e.g., pharmacy) to ensure blinding integrity. Each subject will receive 2 capsules of hyoscine butylbromide or placebo, with a total of 74 bags (or bottles, 2 capsules per bag or bottle) for 74 subjects. Medication numbers will correspond one-to-one with subject randomization numbers. Subjects who pass screening will be randomly assigned to either the hyoscine butylbromide capsules + endoscopy group (treatment group) or the placebo + endoscopy group (placebo group).
3. Study Medication and Concomitant Treatment The hyoscine butylbromide capsules and placebo used in this study are provided by Guangdong Huanan Pharmaceutical Group Co., Ltd. The dosing regimen is as follows: 30 ± 5 minutes before endoscopy, subjects in the treatment group will take 2 capsules (20 mg) of hyoscine butylbromide, while subjects in the placebo group will take 2 capsules of matching placebo identical in appearance to hyoscine butylbromide capsules.

   Concomitant treatment: During the study period (from screening until 24 hours after endoscopy completion), the use of medications in the same class as hyoscine butylbromide or medications with equivalent antispasmodic effects is prohibited. Other medications are permitted, including preoperative preparation medications and anesthetic agents for painless endoscopy, as well as medications for the treatment of adverse events or underlying diseases. The timing of use shall be determined by the investigator.
4. Endoscopy Procedures Endoscopy procedures should be performed using the same equipment whenever possible and preferably by the same endoscopist. Preoperative preparation for painless endoscopy and procedural protocols shall follow institutional regulations, clinical practice, or relevant clinical practice guidelines.
5. Safety Follow-up (Within 24 Hours After Endoscopy Completion) Within 24 hours after endoscopy completion, subjects shall be followed up (telephone follow-up is acceptable) for safety assessment. Vital signs examination shall be completed again within 1 hour after endoscopy completion. Additional examinations or assessments may be performed if other adverse events or abnormal signs are suspected.

During endoscopy and within 24 hours after completion, subjects shall be followed up (telephone follow-up is acceptable) for Visual Analog Scale (VAS) assessment at the time of maximum pain.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤75 years, regardless of sex;
* Patients scheduled to undergo painless gastrointestinal endoscopy examination or endoscopic surgery, which must include upper gastrointestinal endoscopy;
* Voluntary participation based on the free will of the subject or their legal guardian, with signed informed consent form.

Exclusion Criteria:

* Patients with a history of upper gastrointestinal surgery or colorectal surgery;
* American Society of Anesthesiologists (ASA) classification ≥ Grade III;
* Patients with severe cardiac conditions, including severe arrhythmia, structural heart disease, or other serious cardiac disorders;
* Significant hepatic or renal dysfunction affecting drug metabolism, defined as ALT > 2.5 × ULN, AST > 2.5 × ULN, or Scr > 1.5 × ULN;
* Organic pyloric stenosis, paralytic ileus, or other severe organic gastrointestinal diseases that are unsuitable for painless gastrointestinal endoscopy;
* Patients with suspected gastrointestinal ulcer bleeding or perforation;
* Patients with glaucoma or prostatic hypertrophy;
* Pregnant or lactating women;
* Known hypersensitivity to any component of the study drug;
* Use of medications affecting gastrointestinal motility within 7 days prior to study enrollment;
* Other conditions unsuitable for painless endoscopy procedures;
* Participation in another drug or medical device clinical trial within 30 days prior to study enrollment;
* Patients deemed unsuitable for participation in this clinical study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of gastric peristaltic movements per minute at intraoperative recording points | During endoscopy procedure
  Evaluation method and criteria for gastric peristalsis frequency: A third-party investigator will count the number of peristaltic movements from the endoscopic video recordings. After documenting the results, a statistician will calculate the mean value per minute.

SECONDARY OUTCOMES:
Number of intestinal peristaltic movements per minute at intraoperative recording points | During endoscopy procedure
  Evaluation method and criteria for intestinal peristalsis frequency: A third-party investigator will count the number of peristaltic movements from the endoscopic video recordings. After documenting the results, a statistician will calculate the mean value per minute.
Procedural observation time | During endoscopy procedure
  Defined as the time interval from endoscope insertion to complete withdrawal (recorded separately for upper gastrointestinal endoscopy and colorectal endoscopy).

IPD SHARING:
Plan to Share IPD: No